CLINICAL TRIAL: NCT05562440
Title: The Perspective of Healthy Individuals on Breast Cancer Risk Prediction Report in The Indonesian Population (Perspektif Para Individu Sehat Terhadap Laporan Prediksi Risiko Kanker Payudara)
Brief Title: The Perspective of Healthy Individuals on Breast Cancer Risk Prediction Report In The Indonesian Population
Acronym: PERCEPTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nalagenetics Pte Ltd (Industry)
Collaborators: SJH Initiatives (Unknown); MRCCC Siloam Hospitals Semanggi (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ID-BCRPS-02-20220913
Record Dates: First submitted 2022-09-23; First posted 2022-09-30 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Focus Group Discussion
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Focus Group Discussion on breast cancer risk prediction report (Experimental): Woman population with no breast cancer who received the dummy report result
  Interventions: Other: Focus Group Discussion

INTERVENTIONS:
Other: Focus Group Discussion — Each focus group will consist up to five participants in every session, two sessions each for both low and high risk group. Every FGD sessions will last for 1 to 2 hours and be conducted in Indonesian, and will be recorded. Both groups will be asked the following questions: 1) What is your opinion regarding the clarity of information in the dummy breast cancer risk prediction report?; 2) What is your opinion regarding the completeness of information in the dummy breast cancer risk prediction report?; and 3) What is your impression regarding the results presented in the dummy breast cancer risk prediction report?.

SUMMARY:
In 2016, a meta-analysis showed that DNA-based risk reporting alone does not facilitate behavior change. However, there have been several studies showing that tailoring care plans related to diet may help with adherence to a tailored diet plan.

Risk prediction report displays both Polygenic Risk Score (PRS) and modifiable (non-genetic) risk factors. Overtime, the investigators aim to combine both PRS and modifiable risk factors to have a localized and stronger prediction model for the local population. The risk prediction report is designed to tailor care plans for patients by their physicians or care planner.

Focus groups allow deeper discussions in themes important to guide design of the report. This method has been used in previous similar studies, such as one by Cutting et al to understand physicians' preference in integrating genetic reports into daily practice. Studies also have shown that local adoption of personalized medicine and care is hindered by limited infrastructure of information management and awareness, despite personalized medicine being widely adopted in healthcare systems in developing countries.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Able to give informed consent
3. Aged 25-75 years old
4. Have access to a mobile phone or computer with the Zoom application or a caregiver who is able to assist them with the Zoom application

Exclusion Criteria:

1. Ever diagnosed with breast cancer

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The focus of the study is on breast cancer.
Enrollment: 10 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-02-12 (Actual); Study Completion 2023-02-12 (Actual)

PRIMARY OUTCOMES:
Focus Group Discussions | Immediately after exposure to dummy report
  To qualitatively investigate participants' perceptions and gather their feedbacks on the clarity, completeness, and their impressions towards the breast cancer risk prediction dummy report. FGD will be transcribed and analyzed using thematic analysis method.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel J Haryono, Ph.D., MD, Principal Investigator — SJH Initiatives; Faustina A Agatha, S. Biotek, Study Chair — SJH Initiatives; Fatma Aldila, MPH, Study Chair — Nalagenetics Pte Ltd; Eric A Fernandez, Ph.D., Study Chair — Nalagenetics Pte Ltd; Sabrina G Tanu, B. Sci, Study Chair — Nalagenetics Pte Ltd
Locations (1):
- MRCCC Siloam Hospitals Semanggi, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hollands GJ, French DP, Griffin SJ, Prevost AT, Sutton S, King S, Marteau TM. The impact of communicating genetic risks of disease on risk-reducing health behaviour: systematic review with meta-analysis. BMJ. 2016 Mar 15;352:i1102. doi: 10.1136/bmj.i1102. PMID 26979548
- [Background] Vranceanu M, Pickering C, Filip L, Pralea IE, Sundaram S, Al-Saleh A, Popa DS, Grimaldi KA. A comparison of a ketogenic diet with a LowGI/nutrigenetic diet over 6 months for weight loss and 18-month follow-up. BMC Nutr. 2020 Sep 24;6:53. doi: 10.1186/s40795-020-00370-7. eCollection 2020. PMID 32983551
- [Background] Cutting E, Banchero M, Beitelshees AL, Cimino JJ, Fiol GD, Gurses AP, Hoffman MA, Jeng LJ, Kawamoto K, Kelemen M, Pincus HA, Shuldiner AR, Williams MS, Pollin TI, Overby CL. User-centered design of multi-gene sequencing panel reports for clinicians. J Biomed Inform. 2016 Oct;63:1-10. doi: 10.1016/j.jbi.2016.07.014. Epub 2016 Jul 14. PMID 27423699
- [Background] Chong HY, Allotey PA, Chaiyakunapruk N. Current landscape of personalized medicine adoption and implementation in Southeast Asia. BMC Med Genomics. 2018 Oct 26;11(1):94. doi: 10.1186/s12920-018-0420-4. PMID 30367635
- [Background] Liu J, Ho PJ, Tan THL, Yeoh YS, Chew YJ, Mohamed Riza NK, Khng AJ, Goh SA, Wang Y, Oh HB, Chin CH, Kwek SC, Zhang ZP, Ong DLS, Quek ST, Tan CC, Wee HL, Li J, Iau PTC, Hartman M. BREAst screening Tailored for HEr (BREATHE)-A study protocol on personalised risk-based breast cancer screening programme. PLoS One. 2022 Mar 31;17(3):e0265965. doi: 10.1371/journal.pone.0265965. eCollection 2022. PMID 35358246
- [Background] Ho WK, Tan MM, Mavaddat N, Tai MC, Mariapun S, Li J, Ho PJ, Dennis J, Tyrer JP, Bolla MK, Michailidou K, Wang Q, Kang D, Choi JY, Jamaris S, Shu XO, Yoon SY, Park SK, Kim SW, Shen CY, Yu JC, Tan EY, Chan PMY, Muir K, Lophatananon A, Wu AH, Stram DO, Matsuo K, Ito H, Chan CW, Ngeow J, Yong WS, Lim SH, Lim GH, Kwong A, Chan TL, Tan SM, Seah J, John EM, Kurian AW, Koh WP, Khor CC, Iwasaki M, Yamaji T, Tan KMV, Tan KTB, Spinelli JJ, Aronson KJ, Hasan SN, Rahmat K, Vijayananthan A, Sim X, Pharoah PDP, Zheng W, Dunning AM, Simard J, van Dam RM, Yip CH, Taib NAM, Hartman M, Easton DF, Teo SH, Antoniou AC. European polygenic risk score for prediction of breast cancer shows similar performance in Asian women. Nat Commun. 2020 Jul 31;11(1):3833. doi: 10.1038/s41467-020-17680-w. PMID 32737321